CLINICAL TRIAL: NCT06097481
Title: Refining an Asynchronous Narrative-Based Intervention for Adjusting to Heart Failure Chronic Illness to Advance Behavioral Health Equity
Brief Title: Narrative Intervention for Chronic Illness- Heart Failure Trial (NICI-HF)
Acronym: NICI-HF
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23-0436
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Study will have two arms, intervention and sham control arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know if they are in the intervention or sham control arm. Statisticians will not know arm when assessing outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NICI-HF (Experimental): This arm will receive the NICI-HF intervention with regular emails from a therapist for 3 months.
  Interventions: Behavioral: Narrative Intervention for Chronic Illness-Heart Failure
- Sham control (Placebo Comparator): This arm will receive regular emails with information about heart failure for 3 months.
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Narrative Intervention for Chronic Illness-Heart Failure — The Narrative Intervention for Chronic Illness-Heart Failure includes narrative-based, strengths-based, solution-focused brief therapy, and Unitary Caring Science to improve depression (primary outcome) and anxiety (secondary outcome) for people living with heart failure.
  Arms: NICI-HF
Other: Attention Control — Automated emails at similar time points to the intervention will be sent to participants in this arm. Emails will ask participants to reflect on their illness experience and offer general information about heart failure using standardized handouts from the American Heart Association and Up-To-Date.
  Arms: Sham control

SUMMARY:
The Narrative Intervention for Chronic Illness-Heart Failure (NICI-HF) offers an asynchronous interactive text behavioral health intervention to advance behavioral health equity by facilitating access to care for people adjusting to living with heart failure (HF). The proposed study will recruit up to 70 people living with heart failure. This study will gain insight into living with heart failure and learn if the narrative-based intervention is feasible and acceptable for people living with heart failure. The study has two specific aims:

Aim 1: Evaluate the effects of NICI-HF intervention on standard behavioral outcomes. The study investigators will review depression with the Personal Health Questionnaire-9 (primary) and anxiety with the General Anxiety Disorder-7 (secondary) outcomes, and explore self-care with the Self Care for Heart Failure Index by comparing the sham control (n=30) and NICI-HF intervention (n=30) groups at baseline, three months, and six months.

Aim 2: Refine NICI-HF for feasibility and acceptability to support HF self-care and burdensome symptom management and to increase behavioral health equity by improving proximity to services. The study investigators will use standard implementation domains to tailor the intervention for HF using qualitative semi-structured interviews and mixed methods analysis. The study investigators will refine and manualize the intervention for future R01 testing across chronic illnesses with diverse and marginalized populations and service delivery models.

DETAILED DESCRIPTION:
The Refining an Asynchronous Narrative-Based Intervention for Adjusting to Heart Failure Chronic Illness to Advance Behavioral Health Equity study is a NIH Intervention Stage 1B intervention study design with randomization into two arms: a sham control (SC) and an intervention arm (IA). The study investigators will be recruiting up to 64 participants adjusting to living with heart failure. All participants will be randomized to the SC or IA arms (1:1 randomization). All participants will be asked to complete measurements at baseline (T0), three months (T3), and six months (T6). Measurements at T0 include demographic information, Personal Health Questionnaire-9 item (PHQ9), General Anxiety Disorder-7 item (GAD7), Kansas City Cardiomyopathy Questionnaire (KCCQ), and the Self Care Heart Failure Index (SCHFI). T3 measurements include: PHQ9, GAD7, KCCQ, and SCHFI. Measurements at T6 include: PHQ9, GAD7, SCHFI, KCCQ, and self-reported access to care and healthcare utilization. Measurements will be administered by email link using REDCap (an online database administered by the University of Colorado).

Intervention and sham control groups will receive biweekly text response prompts. The IA will have tailored responses crafted by the social work psychotherapists. The SC group will not have feedback or tailored responses.

Study participants who complete Week 8 will also be asked to participate in a semi-structured interview at T3. The study investigators will integrate both quantitative and qualitative results as a convergent mixed methods analysis study. In the mixed analyses, The study investigators will pay attention to points of integration in the qualitative subsample of the population, patterns of behavioral outcome scores, context, geolocation characteristics, access to care experience; and frequency of self-schema, world-schema, and self-care of illness compared across aims.

ELIGIBILITY:
Inclusion Criteria:

* Dx with Heart Failure, NYHA Class III and IV
* Have an email address and able to check email regularly
* Have a working phone number
* Between the ages of 18-89 years old

Exclusion Criteria:

* Conflicting research study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Personal Health Questionnaire 9 item (PHQ9) | Administered at baseline, 3 months, and 6 months
  The Personal Health Questionnaire 9 item (PHQ9) is a measurement of depression, found to be reliable for people living with heart failure. Scores range from 0-27, with higher scores indicating higher depression levels.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder measurement- 7 item (GAD-7) | Administered at baseline, 3 months, and 6 months
  The Generalized Anxiety Disorder measurement- 7 item (GAD-7) is a measurement of anxiety found to be reliable for people living with chronic illnesses like heart failure. Scores range from 0-21 with higher scores indicating higher levels of anxiety.

OTHER OUTCOMES:
Self Care Heart Failure Index (SCHFI) | Administered at baseline, 3 months, and 6 months
  The Self Care Heart Failure Index (SCHFI) is a measurement of heart failure self-care and has been found to be reliable for people living with heart failure. Scores vary from 0-100. A score of 70 or greater can be used as the cut-point to judge self-care adequacy, although evidence is provided that benefit occurs at even lower levels of self-care.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Administered at baseline, 3 months, and 6 months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a self reported heart failure severity measure. Scores range from 0-100: frequently summarized as 25-point ranges with 0 being very poor and 100 being excellent.

IPD SHARING:
Plan to Share IPD: No